CLINICAL TRIAL: NCT03019601
Title: Enhancing Uptake of Family Planning Services by HIV Infected Women Attending the Postpartum Component of the PMTCT Program in Mulago National Referral Hospital, Kampala, Uganda Utilizing HIV-Infected Peers as Family Planning Champions
Brief Title: Enhancing Uptake of Family Planning Services by HIV-Infected Women Attending the PMTCT Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: MU-JHU CARE (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NA_00048133; UM1AI069530 (NIH)
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Contraception
Keywords: HIV; PMTCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group education (Experimental): Non pregnant HIV+ mothers were exposed to a structured educational intervention on family planning facilitated by Peer Champions.
  Interventions: Behavioral: Group Education

INTERVENTIONS:
Behavioral: Group Education — Structured group education on family planning facilitated by Peer Champions

SUMMARY:
A specific organized program utilizing peers in the PMTCT clinic who provide family planning information and support to HIV infected mothers was compared to providing standard family planning messages currently used in the clinic.

DETAILED DESCRIPTION:
A planned group education structural intervention utilizing peers in the PMTCT clinic who provide family planning information and support to HIV infected mothers was compared to the standard of care which consisted of providing standard family planning messages to women attending the PMTCT Clinic. The study had two phases.

The Formative Phase consisted of six focus group discussions and six in depth interviews.

In the Implementation Phase, patient attendance and family planning uptake summaries for during implementation were monitored and summarized daily. Weekly average summaries were considered as time points.

ELIGIBILITY:
Inclusion Criteria:

* This being a program based intervention, all HIV positive mothers who utilize the PMTCT and post natal clinic during the study period will be enrolled.

Exclusion Criteria:

* none

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3300 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
proportion of mothers who took up Family Planning | weekly for one year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mudiope, MBChB, MSc, Principal Investigator — MU-JHU CARE

IPD SHARING:
Plan to Share IPD: No